CLINICAL TRIAL: NCT02837250
Title: Pilot RCT of Patient Centered eHealth Intervention for Nonadherent HIV+ Substance Users
Brief Title: Pilot RCT of Pos4Health for Nonadherent HIV+ Substance Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Ingersoll, PI, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18938; R34DA039011-01 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Nonadherence
Keywords: HIV; Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pos4Health (Experimental): Pos4Health is a 6 Core Internet intervention focusing on improving adherence to ART among nonadherent substance users living with HIV in non urban areas. Pos4Health Cores each present a topic, show videos of HIV+ peers discussing that topic, and how they have coped with it, and use interactions to teach about the topic and to develop knowledge and skills. Each core ends with tips to try that include tips mentioned by peers or from expert material. Content is personalized to the user and users receive tailored feedback. Cores are metered out weekly after each Core is completed.
  Interventions: Behavioral: Pos4Health
- Patient Education (Active Comparator): Patient Education is a static (unchanging) website that presents accurate information about the same topics in Pos4Health, but without personalization, peer videos, or interactivity.
  Interventions: Behavioral: Patient Education

INTERVENTIONS:
Behavioral: Pos4Health — This is a personalized, interactive, patient-centered Internet intervention targeting nonadherence to ART among substance users living with HIV.
  Arms: Pos4Health
Behavioral: Patient Education — This is a patient education website with content about nonadherence to ART pertinent to substance users living with HIV.
  Arms: Patient Education

SUMMARY:
This project has developed a patient-centered eHealth intervention; specifically, an Internet intervention, targeting multiple issues and nonadherence in HIV. The intervention, Pos4Health, includes peer role model videos and evidence-based interactions to promote understanding, coping with, and managing risk factors for nonadherence to ART, and to improve nonadherence itself. In this Pilot Trial, investigators will test the eHealth intervention Pos4Health with PLWH who reside outside urban centers. The pilot trial will determine the acceptability and feasibility of Pos4Health and explore data on HIV clinical outcomes.

DETAILED DESCRIPTION:
Improving treatment adherence among active substance users requires addressing many health barriers beyond substance use alone.(Dr N. Zaller Ph. D, Gillani, & Rich, 2007; Simoni, Amico, Pearson, & Malow, 2008; Willenbring, 2005) Behaviors like smoking and drug use, and experiences like poverty, poor social support, stigma, fear of HIV disclosure, depression, and anxiety, all reduce antiretroviral (ART) adherence and engagement in care, while accelerating disease progression.(Atkinson & Petrozzino, 2009; Bouhnik et al., 2002; Hendershot, Stoner, Pantalone, & Simoni, 2009; Mugavero et al., 2009; Shuter & Bernstein, 2008; Simoni, Frick, & Huang, 2006; Tucker, Burnam, Sherbourne, Kung, & Gifford, 2003; Villes et al., 2007) Improving multiple health behaviors that are related to nonadherence is a promising approach that will be used in the current project. Emerging evidence supports simultaneously targeting multiple health behaviors.(Prochaska et al., 2008) Unfortunately, few interventions address the range of issues that undermine adherence to HIV care.

Extending a program of research by the investigative team, this project will develop a patient-centered eHealth intervention; specifically, an Internet intervention, targeting multiple issues and nonadherence in HIV.

The specific aims are:

1. To develop a prototype of a patient-centered eHealth (Internet) intervention targeting adherence and a set of behaviors and experiences known to undermine adherence among non-urban PLWH.
2. To evaluate the prototype for usability, feasibility and acceptability among PLWH and HIV care clinicians, modify it using PLWH and clinician feedback, and finalize it for pilot testing
3. To pilot test the finalized intervention to determine whether it warrants a subsequent randomized clinical trial.

The pilot test will:

1. evaluate the feasibility of the eHealth intervention by examining access, usage, refusal vs. enrollment, retention vs. dropout, etc. using both web-tracked process data and interviews
2. provide preliminary data on the impact of the eHealth intervention on knowledge and usage of strategies of adherence and each targeted experience and behavior that undermines ART adherence
3. test variables likely to be used as primary outcome markers in a subsequent RCT for their variance in this population (i.e., adherence by pharmacy refill rate, rate of missed HIV care visits, rate of drug-using days, and rate of risky drinking days)

If the pilot test of the new patient-centered eHealth intervention shows an impact on knowledge and use of strategies, and it proves to be feasible and acceptable, it will be tested in a subsequent RCT.

ELIGIBILITY:
Inclusion Criteria:

HIV positive and on ART

* Reports ART nonadherence in the past 30 days (Subject reports missed taking HIV medication at least 5/90 days on the 90 day TLFB at enrollment)
* Screens positive for substance use in the past 30 days (Subject reports using illicit drug at least once on the 90 day TLFB at enrollment) OR Screens positive for alcohol abuse in past 30 days (Subject reports binging or exceeding weekly drinking limit (for women 8 drinks/week; for men 15 drinks/week) at least twice on the 90 day TLFB at enrollment)
* At least 18 years old
* Speaks and reads English
* Can provide meaningful informed consent
* Willing to be followed for 4-5 months
* Has regular access to a phone, email, and computer connected to the Internet

Exclusion Criteria:

* • Never missed an ART dose in past 90 days

  * Reports no use of illicit drugs or risky drinking in past 90 days
  * Cognitive disorders including mental retardation and dementia that could impair ability to understand the intervention material or give informed consent, or psychotic disorder due to the same issues
  * A prisoner, hospitalized, or institutionalized
  * Illiterate
  * Does not have email or ability to access the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Study Acceptance will be determined by consents obtained divided by patients approached for the study. The trial will be considered feasible if the acceptance rate among eligible patients is equal to or greater than 56%.
Acceptability | 6 months
  Is the intervention acceptable? Acceptability will be judged by participant ratings, and by actual program usage data. Participants will rate the Intervention at follow-up. The range of items on this scale is from 1 to 7. An item mean of 3.5 would be mid-range. Basic descriptive information will be gathered from the tracking system about whether participants logged in, how many times, and for how long. Time spent in each Core will be tracked and summarized. Pos4Health will be judged acceptable if if the average score on the evaluation was > 5.6, which is 80% of the highest score (range 1-7), and if 75% of participants completed at least half of the Cores and provide 4 of 7daily diaries of adherence on at least 4 weeks.
Knowledge and Usage of Coping Strategies | 6 months
  The study will compare the Pos4Health and PtEd groups are knowledge and usage of evidence-based coping strategies for the problems targeted by each Core. Linear models will compare change between groups from baseline to post-treatment follow-up.

SECONDARY OUTCOMES:
Adherence by Pharmacy Refill Rate and Treatment Engagement by Missed Visit Proportion | 6 months
  There is 1 secondary research question: How do adherence and engagement in care measures perform as future primary outcomes? Unfortunately, the quantity and quality of adherence and engagement in care indicators (Pharmacy Refill Rate, Missed Visit Proportion) were not adequate to determine which ones are suitable as outcome measures in a future RCT. Our team had hoped to calculate effect sizes for a subsequent randomized trial.

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Ingersoll, Ph.D., Principal Investigator — University of Virginia; Interest Site, Study Director — www.pos4health.org
Locations (1):
- University of Virginia Center for Behavioral Health and Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modipane MB, Waldman AL, Ritterband L, Dillingham R, Bullock L, Ingersoll KS. Technology Use Among Patients in a Nonurban Southern U.S. HIV Clinic in 2015. Telemed J E Health. 2016 Nov;22(11):965-968. doi: 10.1089/tmj.2015.0242. Epub 2016 Apr 28. PMID 27123688

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT02837250/SAP_000.pdf
  • Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT02837250/ICF_001.pdf